CLINICAL TRIAL: NCT01110733
Title: Prospective, Longitudinal, Multinational Registry of Patients With Newly Diagnosed Peripheral T-Cell Lymphoma
Brief Title: Comprehensive Oncology Measures for Peripheral T-cell Lymphoma Treatment Registry
Acronym: COMPLETE
Status: Completed | Type: Observational
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COMPLETE Registry
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Non-Hodgkins Lymphoma; Non-Hodgkin's Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Prospective, longitudinal, multinational, observational study that will collect data on how patients with peripheral T-cell lymphoma (PTCL) are treated in academic and community practices.

DETAILED DESCRIPTION:
The COMPLETE registry is a prospective, longitudinal, multinational, observational study that will collect data on how patients with peripheral T-cell lymphoma (PTCL) are treated in academic and community practices. The registry will enroll newly-diagnosed patients with PTCL treated with a variety of regimens. The COMPLETE registry is designed to better understand PTCL patient characteristics, treatments, and outcomes to help design and understand future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient is newly diagnosed with Peripheral T-cell Lymphoma (PTCL):

  * Aggressive natural killer (NK)-cell leukemia
  * Adult T-cell lymphoma/leukemia (human T-cell leukemia virus [HTLV] 1+)
  * Angioimmunoblastic T-cell lymphoma
  * Anaplastic large cell lymphoma (ALCL), primary systemic type (ALK+, ALK-)
  * PTCL, not otherwise specified (NOS)
  * T/NK-cell lymphoma, nasal type
  * Enteropathy-type intestinal lymphoma
  * Hepatosplenic T-cell lymphoma
  * Subcutaneous panniculitis T-cell lymphoma
  * Transformed mycosis fungoides (at diagnosis of transformation)
  * T-cell prolymphocytic leukemia (T-PLL)
  * Cutaneous gamma/delta (γ/δ) T-cell lymphoma
  * Cutaneous aggressive CD8+ T-cell lymphoma
  * Hematodermic neoplasms (blastic plasmacytoid dendritic cell neoplasm)
  * Systemic Epstein Barr Virus (EBV)+ T-cell lymphomas (T-cell lymphoproliferative disorders of childhood)
  * Other T-Cell lymphomas that are not listed in the Exclusion Criteria
* Patient gives written informed consent

Exclusion Criteria:

* Patient has other T- or NK-cell malignancies including:

  * Precursor T/NK neoplasms
  * T-cell large granular lymphocytic leukemia
  * Mycosis fungoides, other than transformed mycosis fungoides
  * Sézary syndrome
  * Primary cutaneous CD30+ disorders: ALCL and lymphomatoid papulosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be enrolled from academic and community cancer centers in the United States, France, Germany, Italy and Japan.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, MD, Study Chair — Yale University
Locations (68):
- United States (68):
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Moores Cancer Center UCSD, La Jolla, California
  - Wilshire Oncology Medical Group, La Verne, California
  - UCLA, Los Angeles, California
  - USC & Norris Cancer Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - UCLA Olive View Medical Center, Sylmar, California
  - Danbury Hospital Praxair Cancer Center, Danbury, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - Coral Springs Oncology, Coral Springs, Florida
  - Medical Specialists of the Palm Beaches, Lake Worth, Florida
  - Hematology Oncology Associates, Loxahatchee Groves, Florida
  - University of Miami, Miami, Florida
  - MD Anderson Orlando, Orlando, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Emory University Cancer Center, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - UIC Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Simmons Cooper Cancer Institute at SIU School of Medicine, Springfield, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - St. Francis Medical Group Oncology and Hematology Associates, Indianapolis, Indiana
  - Louisiana State University Health Science Center (LSUHSC), Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - ProMedica, Lambertville, Michigan
  - Metro Minnesota Community Clinical Oncology Program, Saint Louis Park, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - St. Louis University Cancer Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital and Morristown Memorial Hospital, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York University Clinical Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center Northeast, Concord, North Carolina
  - Carolina Cancer Management, Inc., Fayetteville, North Carolina
  - Community Cancer Center, Lorain, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - JPS Center for Cancer Care, Fort Worth, Texas
  - South Texas Oncology and Hematology, P.A., San Antonio, Texas
  - Tyler Hematology Oncology, PA, Tyler, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin